CLINICAL TRIAL: NCT04543097
Title: Work And Vocational advicE (WAVE) in Primary Care: a Randomised Controlled Trial
Brief Title: Work And Vocational advicE Study - Effectiveness of Adding a Brief Vocational Support Intervention to Usual Primary Care
Acronym: WAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keele University (Other)
Collaborators: University of Southampton (Other); Guy's and St Thomas' NHS Foundation Trust (Other); University of Birmingham (Other); Aston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RG-0283-19; HTA 17/94/49 (Other Grant/Funding Number: NIHR Health Technology Grant)
Record Dates: First submitted 2020-08-12; First posted 2020-09-09 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Musculoskeletal Pain; Mental Health Issue; Mental Health Disorder; Other Physical Health Condition; Absence
Keywords: Work absence; Other health conditions; Return to work; Musculoskeletal pain; Mental health
MeSH Terms: conditions — Musculoskeletal Pain; Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants, their treating clinicians and VSWs cannot be blinded to allocation due to the nature of the intervention. The data will be analysed independently by two statisticians one of whom will be blinded to intervention allocation the other statistician will be unblinded to allow intervention delivery details to be reported to the Trial Steering Committee (TSC) / Data Monitoring Committee (DMC) if required.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (No Intervention): Participants randomised to the usual care arm will continue to receive care as usual for their health and vocational needs. For most patients, this will comprise usual clinical care, without formal vocational advice.
- Usual care plus vocational support (Experimental): Vocational support following a stepped care model based on the principles of case management in addition to usual primary care.
  Interventions: Behavioral: Vocational Support

INTERVENTIONS:
Behavioral: Vocational Support — Participants randomised to receive vocational advice will all be offered:
  Step 1, contact by phone to undertake an assessment with a trained Vocational Support Worker (VSW) to identify obstacles to Return to Work (RTW) and support RTW planning.
  Step 2, face-to-face (in person or by videoconference) in-depth discussion of obstacles to RTW and further support for RTW planning.
  Step 3, contact by the VSW (with participant consent) with the participants' workplace.
  The frequency of contact will be individualised to the needs of participants and the offer of support continued until sustained RTW (defined as return to any work for at least 4 weeks) or until 6 months of absence, after which participants will be signposted to other services.
  Arms: Usual care plus vocational support

SUMMARY:
Maintaining the population's fitness for work is a priority for the UK Government. People with poor health often struggle at work and take sick leave. Work brings financial, social and health benefits. Few employees receive support to manage their health at work, known as vocational advice, so when their health affects work they visit their general practitioner (GP). The investigators have recently shown the benefits of providing vocational advice for adults consulting in primary care with musculoskeletal pain.

The WAVE study research question is: in patients consulting in general practice who receive a fit note for time off work, does a brief vocational advice intervention lead to fewer days lost from work than usual primary care, and is it cost-effective?

WAVE includes a feasibility phase to adapt a vocational advice intervention for a broader group of patients and test it in a small sample of patients; followed by a pragmatic, multi-centre, two-arm, parallel-group randomised (1:1) trial with internal pilot phase, mixed methods process evaluation and health economic analysis.

Patients will be randomised to either (i) vocational advice intervention plus usual care, or (ii) usual care alone. The vocational advice intervention is designed as a stepped care model based on the principles of case management and delivered by trained Vocational Support Workers (VSWs).

The investigators will also interview patients, General Practitioners (GPs), VSWs and employers to understand their views about the intervention and return to work.

Participants in the trial will be followed-up over 6 months with fortnightly text messages and postal questionnaires at 6 weeks and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and over
* currently in paid employment (full or part time)
* current absence from work of at least two consecutive calendar weeks but not more than six continuous months
* received a fit note
* access to a mobile phone that can receive and respond to SMS text messages
* able to read and write English
* able to give full informed consent
* willing to participate.

Exclusion Criteria:

* Long-term work absence defined as over six continuous months
* pregnancy or on maternity leave
* patients presenting with signs or symptoms indicative of serious illness requiring urgent medical attention ('red' flags)
* severe mental health problems (e.g. severe depression with risk of self-harm, exacerbation of schizophrenia or bipolar disorder, cognitive impairment or lack of capacity)
* high vulnerability (e.g. palliative stages of illness, recent bereavement, dementia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Number of days absent from work | 6 months
  Self reported work absence calculated as the number of days off work over the previous 6 months (since randomisation).

SECONDARY OUTCOMES:
Return to work | 6 months or until sustained return to work (return to any work for 4 consecutive weeks)
  RTW - Self reported number of days until return to work over 6 months, or until a sustained return to work is achieved (defined as return to any work for 4 consecutive weeks).
Work interference | 6 months
  Work Productivity Activity Impairment (WPAI) Questionnaire to measure impairments to work and activities in the past seven days. The WPAI provides four sets of scores; absenteeism, presenteeism, work productivity loss and activity impairment. Scores are multiplied by 100 to express percentages with higher numbers indicating greater impairment and less productivity i.e. worse outcomes.
Work performance | 6 months
  Single Item Productivity Questionnaire (SIPQ) measured using a Visual Analogue Scale with scores ranging from 0 (health has not impacted on work performance at all) to 10 (health is so bad participant has been unable to do their job) a higher score indicates a worse outcome. The scores will be reported as a percentage perceived loss in productivity.

CONTACTS AND LOCATIONS:
Overall Officials: Gwenllian Wynne-Jones, PhD, Principal Investigator — Keele University
Locations (1):
- Keele University, Newcastle-under-Lyme, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Any requests for access to the data from anyone outside of the research team (e.g. collaboration, joint publication, data sharing requests from publishers) will follow the Keele University's data sharing procedure.

REFERENCES:
- [Derived] Wynne-Jones G, Sowden G, Madan I, Walker-Bone K, Chew-Graham C, Saunders B, Lewis M, Bromley K, Jowett S, Parsons V, Mansell G, Cooke K, Lawton SA, Linaker C, Pemberton J, Cooper C, Foster NE. Can vocational advice be delivered in primary care? The Work And Vocational advicE (WAVE) mixed method single arm feasibility study. BMJ Open. 2025 Dec 29;15(12):e098768. doi: 10.1136/bmjopen-2025-098768. PMID 41469060
- See also: Protocol for the Work And Vocational advicE (WAVE) randomised controlled trial testing the addition of vocational advice to usual primary care (Clinical Trials: NCT04543097) — https://doi.org/10.1101/2024.09.11.24313466